CLINICAL TRIAL: NCT00235885
Title: Safety and Efficacy of Adalimumab in Patients With Active Psoriatic Arthritis (PsA) - An Open-Label, Multinational Study to Evaluate the Response to Every-Other Week Adalimumab When Added to Insufficient Standard Therapy, Including Patients Who Failed Prior Treatment With Other TNF-Inhibitors (STEREO)
Brief Title: Safety and Efficacy Study of Adalimumab in Patients With Active Psoriatic Arthritis (PsA)
Acronym: STEREO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M04-724; EudraCT: 2005/001185-14
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; adalimumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

INTERVENTIONS:
Drug: adalimumab

SUMMARY:
The purpose of the study is to assess the safety and clinical efficacy of adalimumab in active psoriatic arthritis (PsA) subjects when adalimumab is added to insufficient standard therapy including patients that have failed other TNF therapies

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age
* Active PsA with > 3 tender and > 3 swollen joints despite standard therapy
* Unsatisfactory response or intolerance to at least one prior or ongoing DMARD (study enrollment must be in accordance with current national guidelines for treatment of PsA with TNF inhibitors)
* A negative serum pregnancy test (serum HCG) for women of childbearing potential prior to the start of treatment.
* Use of a reliable method of contraception by all female patients of childbearing potential
* Able and willing to self-administer sc injections or have a suitable person to administer sc injections
* Able and willing to give written informed consent and comply with the protocol

Exclusion Criteria:

* Prior treatment with any investigational agent within 30 days or five half lives of the product, whichever is longer
* Treatment within last 2 months with infliximab or within last 3 weeks with etanercept
* Treatment within last 4 weeks with a combination of MTX and leflunomide
* Treatment within last 4 weeks with a combination of cyclosporine with any other DMARD-Subject has received UVA phototherapy (including PUVA within 2 weeks prior to screening)
* History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma of the skin or cervical dysplasia
* History of or current active acute inflammatory joint disease of origin other than PsA
* Comorbidities (uncontrolled diabetes, unstable ischemic heart disease, CHF, active IBD, stroke within 3 months, chronic leg ulcer and other condition which would put subject at risk by participation in the protocol
* Positive serology for hepatitis B or C
* History of positive HIV status
* Persistent or recurrent infections or severe infections requiring hospitalization or treatment with iv antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment
* Females who are pregnant or breast-feeding
* History of clinically significant drug or alcohol abuse in the last year
* Previous diagnosis or signs of central nervous system demyelinating diseases
* History of tuberculosis, histoplasmosis or listeriosis
* Subjects with latent TB or having other risk factors for activation of latent TB who have not initiated a TB prophylaxis prior to the first adalimumab treatment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445
Dates: Start 2005-07

PRIMARY OUTCOMES:
Safety parameters
PsARC
ACR20
Physician Global Assessment for Psoriasis and Psoriasis Target Lesion Assessment
Patient reported outcomes

SECONDARY OUTCOMES:
No differentiation will be made between primary and secondary efficacy variables.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Van den Bosch F, Kavanaugh A, Kron M, Kupper H, Mease PJ. Clinical remission in patients with active psoriatic arthritis treated with adalimumab and correlations in joint and skin manifestations. J Rheumatol. 2015 Jun;42(6):952-9. doi: 10.3899/jrheum.140312. Epub 2015 Apr 1. PMID 25834212
- [Derived] Rudwaleit M, Van den Bosch F, Kron M, Kary S, Kupper H. Effectiveness and safety of adalimumab in patients with ankylosing spondylitis or psoriatic arthritis and history of anti-tumor necrosis factor therapy. Arthritis Res Ther. 2010;12(3):R117. doi: 10.1186/ar3054. Epub 2010 Jun 16. PMID 20553600